CLINICAL TRIAL: NCT03511170
Title: A Randomized, Open, Controlled, Multicenter,Phase II Clinical Trial of XELOX and XELIRI Alternative Regimen as First-line Treatment for Advanced Colorectal Cancer
Brief Title: XELOX and XELIRI Alternative Regimen as First-line Treatment for Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harbin Medical University (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Fudan University (Other); Sun Yat-sen University (Other); First Affiliated Hospital of Harbin Medical University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Liaoning Cancer Hospital & Institute (Other); Shengjing Hospital (Other); The First Hospital of Jilin University (Other); The First Affiliated Hospital of Dalian Medical University (Other); Jilin Provincial Tumor Hospital (Other); Jinzhou Medical University (Other)
Responsible Party: Principal Investigator, Yu Han, Chief physician, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-50-IIT
Record Dates: First submitted 2018-04-18; First posted 2018-04-27 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Colorectal Neoplasms; Chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- alternative regiment (Experimental): The first stage:XELOX chemotherapy and XELIRI chemotherapy (alternation of every two cycles) until one of the schemes appears imaging progress or intolerance.And then enter the second stage. The second stage: continue to apply another plan until there is progress or intolerance.
  Interventions: Drug: XELIRI; Drug: XELOX
- classical regiment (Placebo Comparator): Use the XELOX chemotherapy until appears imaging progress or intolerance.And then change to the XELIRI chemotherapy until there is progress or intolerance.
  Interventions: Drug: XELIRI; Drug: XELOX

INTERVENTIONS:
Drug: XELIRI — Irinotecan，200mg/㎡,d1;Capecitabine, 850-1250mg/㎡ bid 1-14;every 21 days as a cycle
Drug: XELOX — Oxaliplatin ,130mg/㎡,d1;Capecitabine, 1000mg/㎡ bid 1-14;every 21 days as a cycle

SUMMARY:
Colorectal cancer will be resistant to Chemotherapy drugs after treated for a period of time .In the past, the classical treatment regiment was to change other drug after tumor progressed. In theory, the continuous use of such a drug could shortening the patient's drug resistance time. It has been shown that the alternate use of the two drug combinations is reasonable in clinical. This application can not only further improve the curative effect but also significantly reduce the side effects. So the investigators are going to carry out a prospective phase II clinical study. The control group change to second-line treatment after progression of first-line drugs. The experimental group use the first line and the second line,alternately, for every two cycles. The combination of bevacizumab is a first line development, and the second line can still be used .Objective to compare the clinical value of XELOX and XELIRI alternation regimen in the first-line treatment of advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as colorectal adenocarcinoma by histopathology and/or cytology.
2. Patients could not receive surgical resection.
3. Never received chemotherapy or radiotherapy.
4. According to the RECIST v1.1 guide, at least 1 lesions (never received radiotherapy),accurately measured by computed tomography (CT) or magnetic resonance imaging (MRI) (intravenous contrast agent as the first choice),the longest diameter was more than 10mm (except for the lymph nodes, the short axis of the lymph nodes must be more than 15mm), repeated measurement.
5. Eastern Cooperative Oncology Group Performance Status(ECOG PS):0-1 score
6. The main organs function is normal, which meets the following requirements. (1) Blood routine examination,(no blood transfusion within 14 days).

   1. Hemoglobin(HB)≥90g/L;
   2. Absolute neutrophil count (ANC) ≥1.5×10^9/L;
   3. Blood platelet (PLT)≥80×10^9/L; (2) Biochemical examination should comply with the following criteria:

   <!-- -->

   1. Bilirubin(BIL) <1.5 times of the upper limit of normal value (ULN)
   2. Alanine aminotransferase (ALT) and aspartate aminotransferase(AST)<2.5*ULN (liver metastasis ALT and AST<5*ULN).
   3. Serum Cr≤1*ULN, creatinine clearance rate≥50ml/min(Cockcroft-Gault formula)
7. The expected survival time more than 3 months;
8. The physicians plan to use XELOX chemotherapy or XELIRI chemotherapy.
9. Patients voluntarily joined the study and signed informed consent form(ICF).
10. Childbearing age women must undergo a negative pregnancy test(serum or urine) within 7 days ,and voluntarily adopt appropriate methods for contraception from the period of under observation and within 8 weeks of the last time they are given the drug;As for men, it is necessary to receive surgical sterilization, or agree to adopt appropriate methods for contraception from the period of under observation and within 8 weeks of the last time they are given the drug.

Exclusion Criteria:

1. There is a case of heart disease in any of the following situations. (1)Recent publications have the following heart disease (within 6 months)

   1. Acute coronary artery syndrome
   2. Acute heart failure (grade III or IV of NYHA classification)
   3. Significant ventricular arrhythmia(sustained ventricular tachycardia, ventricular fibrillation and sudden death after resuscitation).

      (2)The New York Heart Association(NYHA) grade of grade III or IV (3)The patients with severe conduction block, and permanent pacemaker is invalid (two degree and three degree atrioventricular block, sinus arrest) (4)Unexplained syncope occurred within 3 months.

      (5)The researchers identified as uncontrol of severe hypertension, or symptomatic hypertension.
2. There are many factors that affect the absorption of oral drugs (such as unable to swallow, nausea and vomiting, chronic diarrhea and intestinal obstruction).
3. ECOG score≥2
4. Abnormal coagulation function (INR>1.5*ULN, Activated Partial Thromboplastin Time (APTT)>1.5*ULN), with bleeding tendency.
5. There is any history of allergy or hypersensitivity in this research's drug or adjuvant.
6. HIV infection and/or active hepatitis B virus infection.
7. Any condition that may damage the safety of patients or the integrity of research data, including serious medical risk factors, physical condition and laboratory abnormality.
8. The high risk population carrying UGT1A1*28 (7/7) *6 (A/A) genotype or simultaneous carrying of the UGT1A1*28 (6/7) *6 (A/G) genotype (the heterozygous genotype) suggests the exclusion of the Irinotecan
9. Pregnant or lactating women;
10. Other conditions which the doctor think not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 22 months
  Adverse events will be evaluated according to NCI CTCAE 4.0
time to failure of strategy（TFS） | 22 months
  time from the beginning of the treatment until appear the following events, including death and implementation.the progress of disease

SECONDARY OUTCOMES:
Objective response rate (ORR) | 22 months
  The proportion of patients whose tumor is reduced to a certain amount and maintain a certain period of time.
Disease control rate(DCR) | 22 months
  The rate of cases of remission and stable disease accounts for the total evaluable cases after treatment
Overall Survival (OS) | 22 months
  overall survival time after the beginning of the treatment
time to failure of strategy（TFS） | 22 months
  time from the second beginning of the treatment until appear the following events, including death and implementation.the progress of disease

CONTACTS AND LOCATIONS:
Locations (1):
- Harbin Medical University, Harbin, Heilongjiang, China